CLINICAL TRIAL: NCT00770900
Title: Prospective, Randomized, Double-blind, Study to Evaluate the Eosinophils Activation Parameters and Phagocyte Function in Patients With Persistent Asthma Treated With Montelukast
Brief Title: Study to Evaluate the Inflammatory Cells Activity in Patients With Persistent Asthma Treated With Montelukast (0476-403)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Vice President of Late Stage Development, Merck Sharp & Dohme Corp
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008_563; MK0476-403
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2010-12-20 (Estimated); Status verified 2010-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Montelukast (Experimental): Asthmatic children and teenagers took montelukast daily.
  Interventions: Drug: montelukast sodium
- Placebo (Placebo Comparator): Placebo to montelukast tablet daily.
  Interventions: Drug: Comparator: placebo comparator

INTERVENTIONS:
Drug: montelukast sodium — Asthmatic children and teenagers took montelukast daily for 12 weeks.
  Children aged 2-5 years took 4mg tablet of montelukast
  Children aged 6-15 years took 5mg tablet of montelukast
  Children >15 years took 10mg tablet of montelukast
  Other Names: Singulair
  Arms: Montelukast
Drug: Comparator: placebo comparator — Asthmatic children and teenagers took Placebo tablet daily for 12 weeks.
  Arms: Placebo

SUMMARY:
Verify if the quantitative parameters of the eosinophils activation and phagocyte system function show a predictive value for clinical response and prognostic in patients with persistent asthma treated with montelukast

ELIGIBILITY:
Inclusion Criteria:

Patients Between 2-18 Years With Persistent Asthma

Exclusion Criteria:

Patients > 18 Years Old And < 2 Years Old

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Verify if the quantitative parameters of the eosinophils activation and phagocyte system function show a predictive value for clinical response and prognostic. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC